CLINICAL TRIAL: NCT05277272
Title: INTO-HLH- Insight Into the Natural History and Treatment Outcomes of Hemophagocytic Lymphohistiocytosis (HLH): A Disease Registry for Patients With HLH
Brief Title: INTO-HLH: A Disease Registry for Patients With Hemophagocytic Lymphohistiocytosis (HLH)
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Sobi, Inc. (Industry); Baylor College of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0821; Sobi.HLH-RWE102 (Other: Sobi, Inc.)
Record Dates: First submitted 2021-12-29; First posted 2022-03-14 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Hemophagocytic Lymphohistiocytoses
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with clinically suspected or confirmed Hemophagocytic Lymphohistiocytosis: Multi-institutional cohort registry of patients with clinically suspected or confirmed Hemophagocytic Lymphohistiocytosis

SUMMARY:
The purpose of this observational study is to collect data on the natural history of disease of patients with Hemophagocytic Lymphohistiocytosis (HLH) including diagnosis, treatments, responses, and outcomes.

DETAILED DESCRIPTION:
Hemophagocytic Lymphohistiocytosis (HLH) is a complex, hyperinflammatory syndrome resulting from the interplay of genetic predisposition and various environmental factors. Despite available treatment options for HLH, approximately 30% of patients do not respond to therapy. Moreover, the standard therapy is constrained by its toxicities, and safer treatments are pursued.

There is an unmet need for a deeper understanding of the natural history, clinical/etiologic diversity, complications, and treatment outcomes of patients with HLH, specifically from North America. The proposed study, a collaboration between Cincinnati Children's Hospital Medical Center (CCHMC), Texas Children's Hospital, and Sobi Inc. aims to establish a robust registry that will enable investigators to better define the natural history of HLH.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically suspected or confirmed HLH, including those meeting the HLH-2004 diagnostic criteria (primary or secondary forms, including malignancy) and other forms of HLH (macrophage activation syndrome [MAS], cytokine release syndrome [CRS], etc.)
* Signed and dated informed consent and assent (adolescents)

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with clinically suspected or confirmed HLH
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-12-31 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Time to HLH diagnosis from the initial presentation | Interval between date of presentation, as defined as the day of appearance of initial HLH symptom, and the date of full HLH diagnosis, as defined by fulfilling the HLH diagnostic criteria, will be measured. Timeframes up to 6 months will be assessed.
  Date of initial presentation and the date of HLH diagnosis as defined by HLH diagnostic criteria (HLH-2004/MAS classification criteria)
Number of patients with an autoimmune disease at the time of HLH diagnosis | Up to 1 month from HLH diagnosis
  Presence of an autoimmune disease at the time of diagnosis (e.g., Systemic juvenile idiopathic arthritis, lupus)
Number of patients with malignancy at the time of HLH diagnosis | Up to 1 month from HLH diagnosis.
  Presence of hematologic and solid malignancies at the time of HLH diagnosis.
Number of patients treated with immune-activating agents before HLH diagnosis | Up to 1 month before HLH diagnosis.
  The number of patients treated with immune-activating agents before initial diagnosis (checkpoint inhibitors, CAR-T constructs)
Number of patients with central nervous system (CNS) involvement during the HLH disease course. | Up to 1 month from HLH diagnosis.
  CNS involvement as defined by elevated neopterin, white blood cells, or protein at a cerebrospinal fluid or changes in MRI
Frequency of a genetic diagnosis underlying the HLH. | Up to 1 month from HLH diagnosis.
  Data on genetic testing will be gathered and investigators will summarize the number to calculate the frequency of a genetic diagnosis.
Number of patients with infections (e.g., EBV, CMV, HHV6, HIV, fungal, bacterial) at the time of diagnosis. | Up to 1 month from HLH diagnosis.
  The presence of infections at HLH diagnosis (serology and polymerase chain reaction).
Number of patients with organ failure. | Up to 1 year from HLH diagnosis.
  Data will be gathered on organ failure related to HLH (e.g., kidney, lung, CNS).
Number of patients with long-term disease-related complications. | Up to 5 years from HLH diagnosis.
  Data on long-term complications (e.g., impaired growth, impaired cognitive development) will be gathered.

SECONDARY OUTCOMES:
Treatment response rate to HLH-related treatments. | Week two from the start of treatment.
  The response of all treatments for all patients using the criteria used to assess the efficacy of anti-IFN treatment in the NI-0501-04 04 and NI-0501-14 clinical trials.
Time to response to HLH-related therapy for patients in the registry. | Assessed up to 12 weeks from start of treatment.
  The response of all treatments for all patients using the criteria used to assess the efficacy of anti-IFN treatment in the NI-0501-04 04 and NI-0501-14 clinical trials.
The survival probability of patients in the registry | From HLH diagnosis to last follow-up or death, whichever comes first, assessed up to 5 years post-HLH diagnosis.
  Data on the occurrence and date of death and the date of last documentation for living patients will be gathered.
Number of patients who received hematopoietic stem cell transplantation (HSCT) | From HLH diagnoses up to 5 years post-HLH diagnosis.
  Data on the frequency of HSCT will be gathered.
Frequency of hematopoietic stem cell transplantation (HSCT) related complications | From HSCT up to 5 years post HSCT.
  Investigators will gather data on the frequency of primary graft failure and reception of more than one cellular product, secondary graft failure, and chimerism post-HSCT. Primary graft failure is defined as the observed record of failure to achieve an absolute neutrophil count (ANC) of >500/µL by 42 days after HSCT. Secondary graft failure is defined as the observed record of cytopenia after initial engraftment (ANC <500/ µL) and is not related to infection or drug toxicity, loss of donor chimerism <5%. Mixed chimerism is defined as <80% donor cells after day +30.
Number of participants with treatment-related adverse events >/= 3 as assessed by CTCAE 5.0 | From initiation of HLH related treatment up to 30 days following discontinuation of treatment.
  Grade 3 and higher adverse events (per CTCAE 5.0) reported in the medical charts will be collected. The data will be summarized and described using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Jordan, MD, Study Chair — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Data that will be shared include individual participant data that underlie the results reported in the article, after de-identification. Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose. The types of analyses will include research on HLH.
Supporting Information: Study Protocol
Time Frame: Beginning three months and ending 5 years following article publication.
Access Criteria: Proposals should be directed to intohlh@cchmc.org. The requests will be considered by the INTO-HLH steering committee.